CLINICAL TRIAL: NCT01043042
Title: Identification of Inpatients at Risk for Poor Glycemic Control
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 091507
Record Dates: First submitted 2010-01-04; First posted 2010-01-06 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Hypoglycemia; Hyperglycemia
Keywords: hypoglycemia among inpatients; hyperglycemia among inpatients
MeSH Terms: conditions — Hypoglycemia; Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hospitalized patients: patients hospitalized at VUH between 4/1/2008 to 10/31/2009
  Interventions: Other: No interventions will be used in this study

INTERVENTIONS:
Other: No interventions will be used in this study — No interventions will be used in this study

SUMMARY:
Both hypoglycemia and hyperglycemia can be detrimental to hospitalized patients. However, it is not clear which patients are more likely to develop significant problems with hypoglycemia or severe hyperglycemia in the hospital. Our hypothesis is that we will be able to identify risk factors present at admission that identify patients at greater risk of poor inpatient glycemic control

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* hospitalized in VUH

Exclusion Criteria:

* -length of stay < 24 hours
* pregnant women
* patients receiving palliative/hospice care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Candidates for inclusion will include all adult (age ≥ 18 years) patients admitted to Vanderbilt University Medical Center from 04/01/2008 to 10/31/2009. Patients will be excluded if they were pregnant at the time of admission or had length of stay < 24 hours.
Sampling Method: Probability Sample
Enrollment: 33011 (Actual)
Dates: Start 2010-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
hypoglycemia or hypoglycemia | during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Boord, MD MPH, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Hospital, Nashville, Tennessee, United States